CLINICAL TRIAL: NCT06462755
Title: Perioperative Database of Chinese Elderly Patients for Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-R01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients (aged ≥ 65 years): elderly patients undergo surgeries
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
To develop and externally validate a risk prediction model for postoperative acute kidney injury (PO-AKI) in elderly patients undergoing major noncardiac surgery, addressing the current gap in predictive tools for this vulnerable population.

The endpoint was the occurrence of PO-AKI within seven days following surgery. Diagnoses were based on the Kidney Disease: Improving Global Outcomes (KDIGO) criterion. Potential PO-AKI-related perioperative data were retrieved and extracted from electronic medical record for model derivation and validation.

Clinicians may consider implementing this externally validated risk prediction model to stratify elderly patients' PO-AKI risks in the early postoperative phases of noncardiac surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (aged ≥ 65 years) undergoing non-cardiac surgeries

Exclusion Criteria:

* (1) Patients who underwent endoscopic or transplant procedures;
* (2) Patients who underwent surgeries lasting longer than 10 hours;
* (3) Patients who had severe preoperative kidney dysfunction, defined as preoperative sCr levels ≥ 353.6 μmol/L, or a baseline estimated Glomerular Filtration Rate (eGFR) < 15 ml/min per 1.73 m2;
* (4) Patients without sCr values at baseline or during follow-up to detect PO-AKI occurrences.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) undergoing non-cardiac surgeries
Sampling Method: Probability Sample
Enrollment: 57089 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative acute kidney injury | within seven days following surgery
  Postoperative acute kidney injury